CLINICAL TRIAL: NCT02862184
Title: Female Sexual Dysfunction, Risks and Outcomes (FSFI)
Acronym: FSFI
Status: Withdrawn | Type: Observational
Why Stopped: No support staff
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Becky Lynn, MD, Assistant Professor, St. Louis University
Other Study IDs: 26311
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Female Sexual Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many women will likely experience a sexual problem in their lifetimes. The Prevalence of Female Sexual Problems Associated with Distress and Determinants of Treatment Seeking (PRESIDE) study surveyed more than 30,000 U.S. women aged >18 years regarding sexual function. Results from this study estimated that 12% of women experience a diagnosable sexual disorder that causes personal distress, with lack of sexual desire being the most prevalent. - See more at: http://www.uspharmacist.com/content/d/featured_articles/c/56908/#sthash.LTDkyRlR.dpuf

DETAILED DESCRIPTION:
Standard of care includes completion of a sexual dysfunctional questionnaire at every visit. This study will collect information from the questionnaires and office visit and follow the patient for outcomes of successful or non successful treatment.

The purpose of this study is to collect and analyze data on the characteristics of women who present with sexual dysfunction, to evaluate what risk factors contribute to sexual dysfunction and to evaluate what factors contribute to successful treatment of sexual dysfunction.

Upon a visit to the office participants will complete the Female Sexual Function Index (FSFI), this is standard of care for all patients. Research related procedures include: Review of questionnaires and collecting data from medical records regarding medical history, and treatment outcomes. If a participant does not return to the office for a follow up visit (or final visit) the final questionnaire will be sent by their preference (e-mail, phone, or mail) noted in the consent form.

Participates will also be given the option of participating in a "future storage of data". Future testing will be in the area of female sexual dysfunction. Data will be identified by a code number and only the research staff at Saint Louis University will have access to the data.

ELIGIBILITY:
Inclusion Criteria:

Female 18 to 89 years of age Being treated at the Saint Louis University Clinic for Sexual Dysfunction

Exclusion Criteria:

None

-

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Many women will likely experience a sexual problem in their lifetimes. The Prevalence of Female Sexual Problems Associated with Distress and Determinants of Treatment Seeking (PRESIDE) study surveyed more than 30,000 U.S. women aged >18 years regarding sexual function. Results from this study estimated that 12% of women experience a diagnosable sexual disorder that causes personal distress, with lack of sexual desire being the most prevalent
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of women with similar characteristics | 1 year
  Categorical variables will be expressed as frequencies and percentages. Continuous variables will be expressed as means and standard deviations and/or medians and ranges. Parametric and nonparametric statistical analysis will be conducted based on normality of distributions.

SECONDARY OUTCOMES:
Number of women with history of risk factors contribute to sexual dysfunction | 1 year
  Categorical variables will be expressed as frequencies and percentages. Continuous variables will be expressed as means and standard deviations and/or medians and ranges. Parametric and nonparametric statistical analysis will be conducted based on normality of distributions.
Number of women with successful treatment of sexual dysfunction. | 1 year
  Categorical variables will be expressed as frequencies and percentages. Continuous variables will be expressed as means and standard deviations and/or medians and ranges. Parametric and nonparametric statistical analysis will be conducted based on normality of distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Becky Lynn, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No